CLINICAL TRIAL: NCT06432231
Title: The Effects of Low Glycemic Index Diet on Epileptic Seizure Frequency, Oxidative Stress, Mental Health, and Health-related Quality of Life in Children With Drug-resistant Epilepsy
Brief Title: Effects of Low Glycemic Index Diet in Children With Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Gamze Yurtdaş Depboylu, Associate professor, Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-GAP-SABF-0052
Record Dates: First submitted 2024-05-18; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Ketogenic Diet; Drug Resistant Epilepsy; Oxidative Stress; Quality of Life; Psychological Health
MeSH Terms: conditions — Drug Resistant Epilepsy; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low glycemic index diet treatment (Experimental): Children with drug-resistant epilepsy were treated with a low glycemic index diet for 3 months.
  Interventions: Other: Low glycemic index diet treatment

INTERVENTIONS:
Other: Low glycemic index diet treatment — This study was a non-randomized, single centre, pre/post-intervention study. A low glycemic index diet was prescribed by a dietician for 3 months. LGID treatment consisted of 10% (40-60 g) low glycaemic index (glycaemic index <50) carbohydrate, 20-30% protein and 60-70% lipid
  Other Names: LGID

SUMMARY:
The goal of this clinical trial was to evaluate the effectiveness of a low glycemic index diet (LGID) on seizure frequency, oxidative stress markers and quality of life in children with drug-resistant epilepsy. Based upon the aims, the following hypotheses were tested:

1. LGID reduces seizure frequency in children with drug-resistant epilepsy.
2. LGID improves oxidative parameters in children with drug-resistant epilepsy
3. LGID improves quality of life and mental health in children with drug-resistant epilepsy

Participants were prescribed the LGID for 3 months.At baseline and at outpatient clinic follow-ups at 3 months, anthropometric measurements were taken, the strengths and difficulties questionnaire (SDQ), Pediatric Inventory of Quality of Life (PedsQL) and depression scales were administered and samples for biochemical measurements were collected. Diet compliance was evaluated by food consumption records during monthly follow-up visits (at 1 , 2, and 3 months).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy of a low glycemic index diet on seizure frequency, oxidative stress markers and quality of life in children with drug-resistant epilepsy.This study was a prospective, non-randomized, single centre intervention conducted in children with drug-resistant epilepsy. Low glycemic index diet was started on an out-patient basis. Children and their parents were educated about the diet and the effect of the diet on seizures. Children who were willing to follow the diet were included in the study. The research dietitian conducted interviews with patients and their parents at the beginning of the study to explain the principles of the diet.At baseline and at outpatient clinic follow-ups at 3 months, anthropometric measurements were taken, the strengths and difficulties questionnaire (SDQ), Pediatric Inventory of Quality of Life (PedsQL) and depression scales were administered and samples for biochemical measurements including oxidative stress parameters were collected. A 3-day dietary intake chart kept by the parents was reviewed at each monthly visit to check and reinforce compliance. Parents were asked to record the seizure frequency and severity in a seizure diary.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 4-18,
* being diagnosed with drug-resistant epilepsy,
* having more than one seizure per week,
* not having followed a ketogenic diet before.
* willing to come for regular follow up

Exclusion Criteria:

* children with known or suspected congenital metabolic, chronic, and systemic diseases in which ketogenic diet is contraindicated.
* non-compliance with the diet recommended by the patient and/or parents
* enteral tube or parenteral feeding

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Changes in seizure frequency | Baseline and Month 3
  Seizure diary was kept by parents to records seizure frequency and severity
Concentration of antioxidant and oxidant status | Baseline and Month 3
  Measurement of oxidative stress markers (Total Antioxidant Status (TAS), Total Oxidant Status (TOS))
Concentration of Paraoxonase Enzyme Activity | Baseline and Month 3
  Measurement of Paraoxonase Enzyme Activity (PON-1)
Concentration of Malondialdehyde (MDA) | Baseline and Month 3
  Measurement of Malondialdehyde (MDA)
Changes in quality of life | Baseline and Month 3
  "Pediatric Inventory of Quality of Life" was applied to assess health-related quality of life. A higher score corresponds to a higher health-related quality of life. The score ranges from 0 to 100
Changes in psychosocial problems | Baseline and Month 3
  Psychosocial problems were assessed by the "Strengths and Difficulties Questionnaire".The questionnaire includes 25 questions, some of which question positive and some of which question negative behavioral characteristics. These questions are grouped under 5 sub-headings. These are behavioral problems, attention deficit and hyperactivity, emotional problems, peer problems and social behaviors. Each heading is evaluated in itself with scores that range from 0 to 10 and the sum of the first four headings gives the "total difficulty score". While high scores in social behavior reflect the individual's strengths in the social domain, high scores in the other four domains (behavioral problems, attention deficit and hyperactivity, emotional problems, peer problems) reflect that the problem areas are severe.
Changes in depression level | Baseline and Month 3
  Depression status was assessed by the "Children's Depression Scale".Scores that can be obtained from the scale can vary between 0-54. The cut-off point of the depression scale for children is 19, and high scores indicate a high risk of depression.

SECONDARY OUTCOMES:
Concentration of glucose | Baseline and Month 3
  Measurement of glucose
Concentration of insulin | Baseline and Month 3
  Measurement of insulin
Concentration of liver function tests | Baseline and Month 3
  Measurement of Alanine transaminase (ALT) and Aspartate transaminase (AST)
Changes in lipid profile | Baseline and Month 3
  Measurement of total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), serum triglyceride (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Yurtdaş Depboylu, Çiğli, İ̇zmi̇r, Turkey (Türkiye)